CLINICAL TRIAL: NCT05010746
Title: TVMR With the Innovalve System Trial - Pilot Study in Italy
Acronym: TWIST-PILOT-IT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INVL20-01-IT
Record Dates: First submitted 2021-08-11; First posted 2021-08-18 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Mitral Valve Regurgitation (Degenerative or Functional)
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MV replacement with Innovalve MR system (Experimental): MV replacement with Innovalve MR system
  Interventions: Device: Innovalve TMVR system

INTERVENTIONS:
Device: Innovalve TMVR system — Innovalve TMVR system

SUMMARY:
Study to evaluate the safety and performance of the Innovalve mitral valve replacement system

ELIGIBILITY:
Inclusion Criteria:

* Clinically significant, symptomatic mitral regurgitation
* High risk for open-heart surgery
* Meets anatomical criteria

Exclusion Criteria:

* Unsuitable anatomy
* Patient is inoperable
* EF <30%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-01-24 (Actual); Primary Completion 2024-05-04 (Actual); Study Completion 2029-10-04 (Estimated)

PRIMARY OUTCOMES:
Absence of implant or delivery related serious adverse events at 30 days | 30 days
  Absence of implant or delivery related serious adverse events at 30 days

SECONDARY OUTCOMES:
Technical Success | Procedure
  All of the following must be present: i. Absence of procedural mortality; and ii. Successful access, delivery, and retrieval of the device delivery system; and iii. Successful deployment and correct positioning of the first intended device; and iv. Freedom from emergency surgery or reintervention related to the device or access procedure.
Procedural Success | 30 days
  All of the following must be present:
  I. Deployment of the device
  II. Absence of major device- or procedure-related SAEs, including:
  1. Death
  2. Stroke
  3. Life-threatening bleeding (Mitral Valve Academic Research Consortium [MVARC] definition)
  4. Major vascular complications requiring surgery to repair
  5. Major cardiac structural complications requiring surgery to repair
  6. Stage 2 or 3 acute kidney injury (including new dialysis)
  7. Myocardial infarction or coronary ischemia requiring percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG)
  8. Unexpected cardiogenic shock requiring intensive care unit (ICU) admission and treatments such as ultrafiltration or hemodynamic assist devices, including intra-aortic balloon pumps or left ventricular (LV) or biventricular assist device, or prolonged intubation for > 48 hours.
  9. Any valve-related dysfunction, migration, thrombosis, or other complication requiring surgery or repeat intervention
Device Success | 30 days, 3, 6, 12 months and annually up to 5 years
  All of the following must be present:
  1. Absence of procedural mortality or stroke; and
  2. Proper placement and positioning of the device; and
  3. Freedom from unplanned surgical or interventional procedures related to the device or access procedure; and
  4. Continued intended safety and performance of the device, including:
  5. No evidence of major structural or functional failure
  6. No specific, major device-related technical failure issues and complications
  7. Reduction of MR to either optimal or acceptable levels* without significant mitral stenosis (i.e., post-procedure effective orifice area [EROA] ≥ 1.5 cm2 with transmitral mean gradient < 5 mmHg), no greater than mild (1+) paravalvular leak (PVL), and no hemolysis
Patient Success | 1 year
  All of the following must be present:
  1. Deployment of the device
  2. Patient returned to the pre-procedural setting; and
  3. No rehospitalizations or reinterventions for the underlying condition (e.g., MR, heart failure); and
  4. Improvement from baseline in symptoms (e.g., New York Heart Association [NYHA] Class improvement by ≥ 1 class); and
  5. Improvement from baseline in functional status (e.g., 6-minute walk test/distance [6MWT/D] improvement by ≥ 50 m); and
  6. Improvement from baseline in quality-of-life (e.g., Kansas City Cardiomyopathy Questionnaire [KCCQ-12] improvement by ≥ 10 points)
Change in NYHA Class | 30 days, 3, 6, 12 months and annually up to 5 years
  New York Heart Association (NYHA) functional classification of heart failure is based on how much a patient is limited during physical activity. The rating ranges from Class I-IV. Class I = no limitations of physical activity; Class II = slight limitations of physical activity, ordinary physical activity results in fatigue, palpitation, shortness of breath; Class III = marked limitations of physical activity, less than ordinary activity causes fatigue, palpitation, or shortness of breath; Class IV = unable to carry on any physical activity without discomfort, symptoms of heart failure at rest.
Increase in 6MWD | from baseline to 30 days, 3, 6, 12 months and annually up to 5 years
Quality of life change (KCCQ-12) | from baseline to 30 days, 3, 6, 12 months and annually up to 5 years
  The Kansas City Cardiomyopathy Questionnaire (KCCQ) is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. An overall summary score can be derived from the physical function, symptom (frequency and severity), social function, and quality of life domains. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Reduction in MR grade | from baseline to 30 days, 3, 6, 12 months and annually up to 5 years
Atrial septal defects requiring closure | 30 days, 3, 6, 12 months and annually up to 5 years
Change in Montreal Cognitive Assessment (MoCa) | Discharge and 30 days
  The Montreal Cognitive Assessment is a 30-point test assessing multiple cognitive domains, including short-term memory recall, visuospatial abilities, executive function, attention, concentration, working memory, language, and orientation to time and place. Scores are on a 30-point scale; scores 26 and above indicate normal cognitive function. Lower scores may indicate mild cognitive impairment (scores 19-25), moderate impairment (scores 10-18), or severe impairment (scores less than 10).
Composite of MVARC criteria | 30 days, 3, 6, 12 months and annually up to 5 years
  Number of patients who experience composite endpoint events: death due to any cause, repeat hospitalization due to heart failure, disabling stroke, myocardial infarction, life-threatening major bleeding, acute kidney injury, or specific device-related major technical failure issues and complications.
  b. Repeat hospitalization for heart failure c. Disabling stroke d. Myocardial infarction e. Life-threatening major bleeding f. Acute kidney injury g. Specific device-related major technical failure issues and complications

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Colombo, Prof, Principal Investigator — Humanitas IRCCS
Locations (1):
- Humanitas, Milan, Italy

IPD SHARING:
Plan to Share IPD: No